CLINICAL TRIAL: NCT07303036
Title: Chronobiological Determinants of Gut Microbiome: The Effects of Meal Timing and Eating Frequency
Brief Title: Chronobiological Determinants of Gut Microbiome
Acronym: ChronoNutr
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Ozdemir, Assistant Professor, Hacettepe University
Other Study IDs: GO 23/450
Record Dates: First submitted 2025-12-03; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; chrononutrition; dietary intake
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Morbidly obese: People who are classified as morbidly obese (BMI>40 kg/m2)
- Non-obese: People who are classified as non-obese (BMI<30 kg/m2)

SUMMARY:
The aim of this study is to examine how the number of daily eating occasions and the timing of energy intake influence gut microbiome composition in both morbidly obese and non-obese individuals. The analysis is based on baseline data from a case-control study involving 11 non-obese and 23 morbidly obese adults. Participants were excluded if they were younger than 19 or older than 65 years, had an acute or chronic inflammatory condition, had been diagnosed with an infectious disease, cancer, or alcohol dependence, or had used antibiotics within the three months prior to screening.

DETAILED DESCRIPTION:
This study aimed to investigate how the number of daily eating occasions and the timing of energy intake influence gut microbiome composition in morbidly obese and non-obese adults. This case-control study examined the gut microbiota of 23 morbidly obese individuals (BMI > 40 kg/m²) and 11 non-obese individuals (BMI < 30 kg/m²).

Dietary intake was assessed using 24-hour dietary recall records. From these data, the number of meals, total daily energy intake, and the proportion of energy consumed within specific time intervals (06:00-13:00, 13:00-20:00, and 20:00-06:00) were calculated. Energy intake occurring after 20:00 was defined as nighttime eating.

Participant eligibility required individuals to be between 19 and 65 years of age, free from acute or chronic inflammatory diseases, and without diagnoses of infectious diseases, cancer, or alcohol addiction. Additionally, participants were excluded if they had taken antibiotics within the three months preceding the screening.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 19 to 65 years Morbid obesity (case group) Non-obese status, including lean or pre-obese (control group) Willingness to participate in the study Ability to provide informed consent

Exclusion Criteria:

Age < 26 years or > 60 years Presence of acute or chronic inflammatory diseases Diagnosis of infectious diseases History of cancer Alcohol addiction Use of antibiotics within 3 months prior to screening

Ages: 26 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study Population:
  Participants were recruited into three groups:
  Case group: 23 morbidly obese participants Control group: 11 non-obese participants, including lean (n=5) and pre-obese (n=6)
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Gut microbial profiles of participants | Baseline
  Gut microbial profiles of participants at phylum and sub-phylum levels
Meal frequency of participants | Baseline
  Number of meals consumed per day
Total daily energy intake | Baseline
  Total daily energy intake assessed from dietary data (kcal/day)
Distribution of energy intake by time of day | Baseline
  Percentage of total daily energy intake consumed during predefined time periods of the day (e.g., morning, afternoon, evening, night)

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study does not include a data-sharing plan.